CLINICAL TRIAL: NCT01445210
Title: A Randomized Comparison of Single Injection vs. Continuous Saphenous Nerve Block to Supplement a Continuous Sciatic Nerve Block in Postoperative Pain Treatment After Major Ankle Surgery: Clinical Outcome and Cost Analysis
Brief Title: Saphenous Nerve Block: Single Shot Versus Continuous Infusion to Supplement a Continuous Sciatic Nerve Block After Major Ankle Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011-0184
Record Dates: First submitted 2011-09-29; First posted 2011-10-03 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-10

CONDITIONS: Major Ankle Surgery
Keywords: Postoperative pain; Major ankle surgery; Continuous nerve block; Saphenous nerve; Ropivacaine
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0,2% Ropivacaine (Active Comparator): Patients randomized to the experimental group receive a continuous infusion of 0,2 % Ropivacaine by elastomeric infusion pump at 5 ml/h in the saphenous catheter after major ankle surgery. Infusion for 48 postoperative hours.
  All patients receive a preoperative single shot of Ropivacaine around saphenous and sciatic nerve and a postoperative continuous sciatic nerve block.
  Interventions: Procedure: Continuous saphenous nerve block
- Control (Placebo Comparator): Patients randomized to the control group receive a continuous infusion of isoton saline by elastomeric infusion pump at 5 ml/h in their catheter after major ankle surgery. Infusion for 48 postoperative hours.
  All patients receive a preoperative single shot of Ropivacaine around saphenous and sciatic nerve and a postoperative continuous sciatic nerve block.
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Continuous saphenous nerve block — 0,2% Ropivacaine by elastomeric infusion pump at 5 ml/h for 48 postoperative hours
  Other Names: Naropin
  Arms: 0,2% Ropivacaine
Procedure: Placebo — Isoton saline by elastomeric infusion pump at 5 ml/h for 48 postoperative hours
  Arms: Control

SUMMARY:
The most useful method to manage pain after major ankle surgery is infusion of local analgesics with a catheter close to the sciatic nerve.

Sensation from the ankle are carried by three nerves: The tibial and peroneal nerve (unified in the sciatic nerve) and the saphenous nerve.

Study purpose is to test whether continuous infusion of local analgesics by saphenous nerve catheter provide a better treatment of pain in comparison with a single injection nerve block. In addition cost-effectiveness of the two methods are compared.

The 50 patients of the trial are randomized in clusters of ten. We intend to do a preliminary analysis of the data from the first 40 patients. However, it is not an interim analysis. Fifty patients will be included independent of the result of the preliminary analysis. The random allocation of the last 10 patients will also be double-blinded.

DETAILED DESCRIPTION:
Major ankle surgery are known to be very painful the first 48 hours after the operation due to surgical oedema. This pain is difficult to control with systemic analgesics. Pain relief with systemic analgesics requires high doses of intravenous opioids and is associated with breakthrough pain and adverse effects of opioids (sedation, nausea, vomiting, obstipation, urinary retention, respiratory depression).

Continuous, peripheral nerve block with catheter technique for two days minimizes the need for systemic analgesics. Today such a continuous sciatic nerve block is part of the standard pain treatment after major ankle surgery on Aarhus University Hospital. Despite accurate placement of the catheter many patients are in great pain because the saphenous nerve remain unaffected. A single injection block relieve the pain but a block with Ropivacaine only last 8-15 hours.

Severe postoperative pain leads to high opioid dosages, cognitive blurring, nausea, vomiting, reduced ambulation, increased surgical stress response and increased morbidity. Pain problems and adverse effects prolongs postoperative observation time and maybe also time to discharge.

The aim of the study establish whether continuous saphenous nerve block is efficient (pain relief or reduced opioid consumption) and justified (cost-effectiveness analysis) compared with single injection block.

ELIGIBILITY:
Inclusion Criteria: Elective major ankle surgery

* total ankle arthroplasty
* subtalar fusion
* ankle fusion (non arthroscopic)

Exclusion Criteria:

* coagulation abnormalities
* infection in the region of needle insertion
* systemic infection
* preoperative consumption of high dose opioid
* preoperative sciatic or femoral nerve neuropathy
* preoperative sensory deficit in either of the lower extremities
* Charcot-Marie-Tooth disorder
* diabetic neuropathy
* severe peripheral vascular disease
* allergy to local anesthetics
* lack of understanding of Numeric Rank Scale (NRS)
* communication problems
* dementia
* body mass index above 35
* bilateral continuous sciatic nerve block
* lack of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Accumulated opioid consumption | First 48 hours postoperative

SECONDARY OUTCOMES:
Success rate for saphenous nerve analgesia | Postoperative, first 48 hours
  Pain rated by NRS and opioid consumption
Success rate for clinical analgesia of foot and ankle | Postoperative, first 48 hours
  Pain rated by NRS and opioid consumption
Success rate for tibial and peroneal nerve block | Postoperative, first 48 hours
  Pain rated by NRS and test of sensation on the toes
Localisation of worst pain | Postoperative, first 48 hours
Cost-effectiveness | 2 first postoperative days

CONTACTS AND LOCATIONS:
Overall Officials: Thomas F Bendtsen, ph.d., MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Fisker AK, Iversen BN, Christensen S, Linde F, Nielsen KK, Borglum J, Bendtsen TF. Combined saphenous and sciatic catheters for analgesia after major ankle surgery: a double-blinded randomized controlled trial. Can J Anaesth. 2015 Aug;62(8):875-82. doi: 10.1007/s12630-015-0379-y. Epub 2015 Apr 8. PMID 25851020